CLINICAL TRIAL: NCT06469788
Title: Improving COVID-19 Vaccine Uptake Among Racial and Ethnic Minority Groups With Rheumatic Diseases
Brief Title: Testimonials and Navigation in Rheumatology
Acronym: TANGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Maria Danila, MD, MSc, MSPH, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-300012168; 5R01MD019235 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Rheumatologic Disease; Autoimmune Diseases
Keywords: COVID-19 vaccination; Rheumatic Diseases
MeSH Terms: conditions — Collagen Diseases; Autoimmune Diseases; Rheumatic Diseases | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Storytelling" video including patient narratives, brochure and patient navigation (Experimental): Participants will review video with narratives on COVID-19 vaccination in patients with AIRD, receive brochure on the same topic; and interact with patient navigators.
  Interventions: Behavioral: Video comprised of AIRD patient narratives on COVID-19 vaccination thoughts and experiences; Behavioral: Brochure on COVID-19 vaccination in AIRD patients; Behavioral: Patient Navigation
- Attention Control: "Oral Health" video and "Oral Health" brochure (Active Comparator): Participants will review video on the importance of oral health in patients with AIRD and receive brochure on the same topic.
  Interventions: Behavioral: Video on the importance of good oral health for patients with AIRD; Behavioral: Brochure on the importance of good oral health in AIRD patients

INTERVENTIONS:
Behavioral: Video comprised of AIRD patient narratives on COVID-19 vaccination thoughts and experiences — Participants will watch video focused on the importance of receipt of updated COVID-19 vaccination in patients with AIRD
  Arms: "Storytelling" video including patient narratives, brochure and patient navigation
Behavioral: Video on the importance of good oral health for patients with AIRD — Participants will watch video on the importance of good oral health in AIRD patients.
  Other Names: Attention Control
  Arms: Attention Control: "Oral Health" video and "Oral Health" brochure
Behavioral: Brochure on COVID-19 vaccination in AIRD patients — Participants
  Arms: "Storytelling" video including patient narratives, brochure and patient navigation
Behavioral: Patient Navigation — Participants will receive phone calls from patient navigators to provide support and information for receipt of updated COVID-19 vaccination in patients with AIRD
  Arms: "Storytelling" video including patient narratives, brochure and patient navigation
Behavioral: Brochure on the importance of good oral health in AIRD patients — Participants will receive a brochure on the importance of good oral health in AIRD patients.
  Arms: Attention Control: "Oral Health" video and "Oral Health" brochure

SUMMARY:
The overall goal of this study is to determine whether a novel, multi-modal, patient-directed behavioral intervention initiated in rheumatology clinics is an effective approach to improve uptake of updated COVID-19 vaccine.

DETAILED DESCRIPTION:
Black and Latinx persons are at higher risk for certain autoimmune and inflammatory rheumatic diseases (AIRD) and have experienced worse COVID-19 outcomes compared to their white counterparts. Given the risks of severe COVID-19 outcomes such as hospitalization and death in people with AIRD, COVID-19 vaccine is recommended in this population. Historically, overall vaccine uptake among people with AIRDs has been low, and this vaccine reluctance has extended to COVID-19 vaccination. While additional COVID-19 vaccine doses have offered considerable added protection against severe outcomes, only 20% of all vaccinated persons in Alabama (AL) and 45% in Massachusetts have obtained an additional dose of COVID-19 vaccine as of October 2022. Racial and ethnic minority groups have faced disparities in obtaining subsequent COVID-19 vaccines, particularly in under-resourced communities, including those in Alabama and Massachusetts. Together, these obstacles exacerbate existing health inequities among people of color and perpetuate worse COVID-19 outcomes.

We will conduct a randomized controlled study to test an intervention that seeks to address gaps in COVID-19 vaccine information and access inequities common in Black and Latinx populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years) with known AIRD
* Black race and/or Latinx ethnicity
* Individuals who have not obtained the updated COVID-19 vaccine series (self-report)

Exclusion Criteria:

-Lack of access to phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Receipt of updated COVID-19 vaccination. | 3 months
  We will measure rates of receipt of updated COVID-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Maria I Danila, MD, MSc, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Brigham Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman CH, Ramsey-Goldman R. Widening Disparities Among Patients With Rheumatic Diseases in the COVID-19 Era: An Urgent Call to Action. Arthritis Rheumatol. 2020 Sep;72(9):1409-1411. doi: 10.1002/art.41306. Epub 2020 Aug 9. No abstract available. PMID 32379381
- [Background] Hmamouchi I, Winthrop K, Launay O, Dougados M. Low rate of influenza and pneumococcal vaccine coverage in rheumatoid arthritis: data from the international COMORA cohort. Vaccine. 2015 Mar 17;33(12):1446-52. doi: 10.1016/j.vaccine.2015.01.065. Epub 2015 Feb 7. PMID 25659279
- [Background] Costello R, Winthrop KL, Pye SR, Brown B, Dixon WG. Influenza and Pneumococcal Vaccination Uptake in Patients with Rheumatoid Arthritis Treated with Immunosuppressive Therapy in the UK: A Retrospective Cohort Study Using Data from the Clinical Practice Research Datalink. PLoS One. 2016 Apr 20;11(4):e0153848. doi: 10.1371/journal.pone.0153848. eCollection 2016. PMID 27096429
- [Background] Boucher VG, Pelaez S, Gemme C, Labbe S, Lavoie KL. Understanding factors associated with vaccine uptake and vaccine hesitancy in patients with rheumatoid arthritis: a scoping literature review. Clin Rheumatol. 2021 Feb;40(2):477-489. doi: 10.1007/s10067-020-05059-7. Epub 2020 Jul 3. PMID 32621081
- [Background] Hua C, Morel J, Ardouin E, Ricard E, Foret J, Mathieu S, Combe B, Lukas C. Reasons for non-vaccination in French rheumatoid arthritis and spondyloarthritis patients. Rheumatology (Oxford). 2015 Apr;54(4):748-50. doi: 10.1093/rheumatology/keu531. Epub 2015 Feb 8. No abstract available. PMID 25667433
- [Background] Qendro T, de la Torre ML, Panopalis P, Hazel E, Ward BJ, Colmegna I, Hudson M. Suboptimal Immunization Coverage among Canadian Rheumatology Patients in Routine Clinical Care. J Rheumatol. 2020 May 1;47(5):770-778. doi: 10.3899/jrheum.181376. Epub 2019 Jul 15. PMID 31308211
- [Background] Curtis JR, Johnson SR, Anthony DD, Arasaratnam RJ, Baden LR, Bass AR, Calabrese C, Gravallese EM, Harpaz R, Kroger A, Sadun RE, Turner AS, Williams EA, Mikuls TR. American College of Rheumatology Guidance for COVID-19 Vaccination in Patients With Rheumatic and Musculoskeletal Diseases: Version 3. Arthritis Rheumatol. 2021 Oct;73(10):e60-e75. doi: 10.1002/art.41928. Epub 2021 Aug 4. PMID 34346564
- [Background] Fernandez-Ruiz R, Masson M, Kim MY, Myers B, Haberman RH, Castillo R, Scher JU, Guttmann A, Carlucci PM, Deonaraine KK, Golpanian M, Robins K, Chang M, Belmont HM, Buyon JP, Blazer AD, Saxena A, Izmirly PM; NYU WARCOV Investigators. Leveraging the United States Epicenter to Provide Insights on COVID-19 in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2020 Dec;72(12):1971-1980. doi: 10.1002/art.41450. Epub 2020 Oct 28. PMID 32715660
- [Background] Gianfrancesco MA, Leykina LA, Izadi Z, Taylor T, Sparks JA, Harrison C, Trupin L, Rush S, Schmajuk G, Katz P, Jacobsohn L, Hsu TY, D'Silva KM, Serling-Boyd N, Wallwork R, Todd DJ, Bhana S, Costello W, Grainger R, Hausmann JS, Liew JW, Sirotich E, Sufka P, Wallace ZS, Machado PM, Robinson PC, Yazdany J; COVID-19 Global Rheumatology Alliance. Association of Race and Ethnicity With COVID-19 Outcomes in Rheumatic Disease: Data From the COVID-19 Global Rheumatology Alliance Physician Registry. Arthritis Rheumatol. 2021 Mar;73(3):374-380. doi: 10.1002/art.41567. Epub 2021 Feb 2. PMID 33146001
- [Background] Taylor T, Yazdany J, Gianfrancesco MA. The racial/ethnic and sociocultural aspects of the pandemic in rheumatology. Best Pract Res Clin Rheumatol. 2021 Mar;35(1):101665. doi: 10.1016/j.berh.2021.101665. Epub 2021 Feb 18. PMID 33648855
- [Background] Raiker R, DeYoung C, Pakhchanian H, Ahmed S, Kavadichanda C, Gupta L, Kardes S. Outcomes of COVID-19 in patients with rheumatoid arthritis: A multicenter research network study in the United States. Semin Arthritis Rheum. 2021 Oct;51(5):1057-1066. doi: 10.1016/j.semarthrit.2021.08.010. Epub 2021 Aug 20. PMID 34450504
- [Background] Pablos JL, Galindo M, Carmona L, Lledo A, Retuerto M, Blanco R, Gonzalez-Gay MA, Martinez-Lopez D, Castrejon I, Alvaro-Gracia JM, Fernandez Fernandez D, Mera-Varela A, Manrique-Arija S, Mena Vazquez N, Fernandez-Nebro A; RIER Investigators Group; RIER investigators group. Clinical outcomes of hospitalised patients with COVID-19 and chronic inflammatory and autoimmune rheumatic diseases: a multicentric matched cohort study. Ann Rheum Dis. 2020 Dec;79(12):1544-1549. doi: 10.1136/annrheumdis-2020-218296. Epub 2020 Aug 12. PMID 32796045
- [Background] England BR, Roul P, Yang Y, Kalil AC, Michaud K, Thiele GM, Sauer BC, Baker JF, Mikuls TR. Risk of COVID-19 in Rheumatoid Arthritis: A National Veterans Affairs Matched Cohort Study in At-Risk Individuals. Arthritis Rheumatol. 2021 Dec;73(12):2179-2188. doi: 10.1002/art.41800. Epub 2021 Oct 19. PMID 33955209